CLINICAL TRIAL: NCT07151222
Title: The Red Blood Cell as a Mediator and Therapeutic Target in Cardiovascular Disease
Brief Title: Role of Red Blood Cells in Cardiovascular Disease
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, John Pernow, Professor, Karolinska Institutet
Other Study IDs: 2024-02534
Record Dates: First submitted 2025-02-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus
Keywords: Red blood cells; Nitric oxide; diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Type 2 diabetes: Patients with type 2 diabetes
- Type 1 diabetes: Patients with type 1 diabetes
- Coronary artery disease/Myocardial infarction: Patients with acute coronary syndromes
- Healthy controls: Age- and gender-matched healthy subjects

SUMMARY:
The risk of myocardial infarction is dependent on cardiovascular risk factors including type 2 diabetes (T2D) but underlying mechanisms are poorly understood. We identified that red blood cells (RBCs) mediate beneficial cardiovascular regulatory effects under hypoxic/ischemic conditions via signaling by nitric oxide (NO) and soluble guanylate cyclase (sGC) in the RBCs. The RBCs become dysregulated in T2D which induces endothelial and cardiac injury. This project investigates the signaling of RBCs in cardiovascular disease and explores novel therapeutic strategies that target RBC function in myocardial infarction and T2D.

Aims To determine the

* mechanisms behind cardioprotective effect of RBCs in myocardial infarction
* signaling behind cardiovascular injury induced by RBCs in T2D

Work plan RBCs collected from patients with myocardial infarction, patients with T2D and healthy controls are investigated in bioassays including isolated hearts of ischemia/reperfusion, endothelial function and cell cultures. Molecular mechanisms behind the effects of RBCs are identified with focus on the NO-sGC pathway in the RBCs.

This project unravels the RBC as a mediator of cardiovascular disease and has the potential to identify novel therapeutic strategies by targeting RBC signaling.

DETAILED DESCRIPTION:
The function of RBCs are investigated in functional bioassays and cell culture systems. The bioassays include isolated hearts subjected to ischemia-reperfusion and isolated arteries. the readouts are left ventricular function, infarct size and endothelial function . Comparisons are made between RBCs collected from patients with cardiovascular disease, type 2 diabetes and healthy controls. Pharmacological interventions are performed by ex vivo incubations with focus on the NO-sGC pathway.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes

Exclusion Criteria:

-

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Red blood cell function defined as their ability to modulated post-ischemic recovery of left ventricular developed pressure, myocardial infarct size and endothelium-dependent relaxation. | At 60 min of reperfusion
  The function of red blood cells (RBCs) are investigated in isolated heart preparations and in isolated aorta.
  The heart preparations are subjected to ischemia followed by 60 min reperfusion and RBCs are administered into the coronary circulation at the onset of ischemia. Left ventricular developed pressure is recorded as readout of left ventricular function. Final infarct size is determined at the end of the reperfusion period.
  Isolated arteries are co-incubated with the RBCs for 18 h. Following the incubation, the arteries are mounted in myographs for the determination of endothelium-dependent and endothelium-independent relaxations.

SECONDARY OUTCOMES:
Red blood cell production of reactive oxygen species | At baseline and following ex vivo inhibition of ROS formation.
  Red blood cell (RBC) production of reactive oxygen species (ROS) is determined at baseline and following incubation of the RBCs with pharmacological tools that modulate different sources of ROS formation. These include nitric oxide synthase inhibitors, NADPH-oxidase inhibitors, arginase inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: John Pernow, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Swsden, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pernow J, Yang J. Red blood cells: a new target to prevent cardiovascular disease? Eur Heart J. 2024 Oct 21;45(40):4249-4251. doi: 10.1093/eurheartj/ehae454. No abstract available. PMID 39258963